CLINICAL TRIAL: NCT01101828
Title: Self-collected Swabs for HPV Testing in 18-24 Year Old Women
Acronym: DRY
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Rachel L. Winer/Assistant Professor, University of Washington
Other Study IDs: 37822-A
Record Dates: First submitted 2010-04-07; First posted 2010-04-12 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Self-collected vaginal samples for HPV testing
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare methods for transporting self-collected swabs for HPV testing in 18-24 year old women and to look at risk factors for HPV infection in 18-24 year old women.

DETAILED DESCRIPTION:
We propose a cross-sectional study among 150 women in the United States who have used Internet dating sites in the past year in order to examine risk factors for high-risk HPV infections in 18-24 year old online daters, and evaluate strategies for transporting and storing self-collected samples for HPV testing. We will ask participants to complete a written questionnaire on their health, sexual behavior, and attitudes toward self-collecting vaginal swabs, HPV vaccination, and cervical cancer screening. Also, we will ask the women to self-collect two sequential vaginal swab samples that will be transported and stored according to the two strategies described above. Each sample will be tested for type-specific HPV DNA using a PCR-based assay.

ELIGIBILITY:
Inclusion Criteria:

* Have had sex with men
* Have used the internet to search for romantic partners in the past year (e.g. posted or responded to an ad on an internet dating website or social networking website)

Exclusion Criteria:

* Pregnant or breastfeeding

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18 to 24 year old women who date online
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Presence of type-specific HPV DNA in self-collected vaginal swab samples | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Winer, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- See also: (HPV study website) — http://depts.washington.edu/hhhstudy/hpv/